CLINICAL TRIAL: NCT02780817
Title: Motor Adaptation by Error Augmentation Force Field in Healthy Peoples' Upper Extremity, a Randomized Controlled Trial
Brief Title: Motor Adaptation by Error Augmentation Force Field in Healthy Peoples' Upper Extremity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 036/15
Record Dates: First submitted 2016-02-28; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Error enhancement (Experimental): Arm reaching rehabilitation training with error-augmentation perturbation forces. One session of about 25 minutes of practicing arm reaching movements on 3D robotic device.
  Interventions: Other: Error enhancement
- Control group (Other): Arm reaching rehabilitation training without error-augmentation perturbation forces. One session of about 25 minutes of practicing arm reaching movements on 3D robotic device.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Error enhancement — Participants will sit in front of a 3D robotic device and grab the robotic arm handle. The participants will carry out arm reaching tasks appear on a screen on front of them. Each game of tasks will lasts 2 minutes. The participants will carry out one game to be accustomed to device, followed by one game with null force field, followed by 5 games as the main intervention with error enhancement force field, and another last game with null force field.
  Arms: Error enhancement
Other: Control group — Participants will sit in front of a 3D robotic device and grab the robotic arm handle. The participants will carry out arm reaching tasks appear on a screen on front of them. Each game of tasks will lasts 2 minutes. The participants will carry out one game to be accustomed to device and another 7 games with null force field.
  Arms: Control group

SUMMARY:
Inducing a systematic perturbation forces on the hand during arm reaching movement may improve adaptation. Error-augmentation (EA) training is relatively new concept in motor learning intended to promote the adaptation process. In this study participants will practice one session of training on 3D robotic device. Healthy volunteers will be randomly divided into two groups: study and control. The study group will carry out the training session with EA forces. The control group will carry out the same procedure with null force field. Outcome measure are the average size of trajectory error from the straight line and level of exertion (borg scale).

DETAILED DESCRIPTION:
A single process involved in motor learning is adaptation. Hand reaching movement has been extensively used to evaluate the concept of motor adaptation. By inducing a systematic perturbation on the hand, it is possible to examine the implicit motor response on the trajectory of the hand. Error-augmentation (EA) training is relatively new concept in motor learning intended to promote the adaptation process. Applying these perturbating forces on the hand shift the hand trajectory form the straight line to a curve like shape. Making repetitive movement under the same conditions will results in a gradual correction of this faulty movement trajectory toward the straight line, e.g. motor adaptation.

Participants: Healthy volunteers, aged 20-50, males and females. The participants will be randomly assigned into two groups: study or control group.

Procedure: One practice session of 25 minutes on 3D robotic device. The study group will carry out the session with EA forces. The control group will carry out the same training without the EA forces.

Outcome Measures: Size of trajectory error from the straight line, level of exertion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Neurologic disease, orthopedic syndrome of the dominant upper extremity.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in average movement error from baseline | At baseline, before the beginning of the training session, and at followup measurement immediately at the the end of the training session, which is about 45 minutes after the first evaluation.
  Average size of trajectory error form the straight line while making arm reaching movement

SECONDARY OUTCOMES:
Change in Borg scale score from baseline | At baseline, before the beginning of the training session, and at followup measurement immediately at the end of the training session, which is about 45 minutes after the first evaluation.
  A 6-20 scale that intended describe the subjective level of exertion of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Carmeli, PhD., Principal Investigator — Professor
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Journal article